CLINICAL TRIAL: NCT02553564
Title: A Randomized Controlled Trial of a Checklist Intervention to Reduce 30 Day Rehospitalization Risk in Hemodialysis Patients
Brief Title: 30 Day Rehospitalization Risk in Hemodialysis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment as expected
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Steven Fishbane, Chief, Division of kidney diseass and Hypertension, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nephrology - 06032015
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Re-hospitalization Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Checklist driven clinical encounter after hospital discharge
  - Participant will receive standard medical care with the addition of a checklist driven clinical encounter upon return to the dialysis unit after hospital discharge.
  * participants in both group will be receiving standard post discharge care which includes nursing assessment, social work intervention as needed and new dialysis orders.
  Interventions: Other: Checklist driven clinical encounter after hospital discharge
- Usual care group (No Intervention): Participant will receive standard medical care upon return to the dialysis unit after hospital discharge.
  * participants in both group will be receiving standard post discharge care which includes nursing assessment, social work intervention as needed and new dialysis orders.

INTERVENTIONS:
Other: Checklist driven clinical encounter after hospital discharge — Within 96 hours of hospital discharge an Nurse Practitioner will perform a checklist guided assessment to preventing rehospitalizations. The assessment consists of the following:
  1. The participants's hospital course will be reviewed and their clinical recovery and stability assessed.
  2. Determination of the participants's estimated dry weight (EDW).
  3. The participants's post discharge medications will be checked, compared to the prehospitalization medication, and discrepancies will be reviewed and corrected.
  4. Blood tests will be ordered for the participants's first return dialysis treatment if medically appropriate after clinical assessment.
  5. Write new dialysis orders.
  6. Dialysis Access- review access and determine any changes required in treatment
  Arms: Intervention group

SUMMARY:
After a hospitalization, dialysis patients have a high risk of being admitted to the hospital again within 30 days. The purpose of this research study is to test a new way of reducing the chance of patients being hospitalized again. In this study investigator will evaluate a checklist driven evaluation upon return to the dialysis facility as a method to reduce the rate of rehospitalizations in hemodialysis patients.

DETAILED DESCRIPTION:
There are an excessive number of 30 day readmissions after hospital discharges of dialysis patients in the U.S. (35.2%). Investigators recent research has found that approximately 2/3 of these readmissions are potentially avoidable. Investigators believe that among the causes for the excessive number of readmissions, the most important may be that patients usually do not receive a clinical assessment upon return to dialysis after a hospitalization. An all too common practice in the U.S. is for the nephrologist to not see the patient but to give verbal orders to the dialysis nurse to resume previous orders. This increases readmission risk in that there are a number of key clinical processes that if completed on return to dialysis might greatly reduce rehospitalization risk. Nephrologists are often not available to see patients in the peri-discharge period, but there is a trend towards an increasing number of U.S. dialysis facilities now having nurse practitioners (NP) working in the units. Investigators believe that NPs using a checklist can conduct a post-discharge clinical encounter that would allow for key care processes to be carried out and to direct telephone communication with the treating nephrologist. Our objective is to reduce the risk of dialysis patient readmissions within 30 days through the use of this intervention. Our research question is whether this intervention would be effective for reducing 30 day readmission risk. Our hypothesis is that the intervention will prove to be more effective then usual care for reducing 30 day readmission risk.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must have been an existing patients of the outpatient dialysis units for at least 1 month prior to the index hospitalization
* Index hospitalization must be from an acute care hospital

Exclusion Criteria:

* Hospital discharges against medical advice
* Assessment cannot be initiated within 96 hours of hospital discharge
* Primary hospital diagnosis related to cancer, renal transplant, mental health or rehabilitation
* Hospital admission was the 5th or more in the previous 12 months
* Failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Rehospitalization rate | Up to 5 weeks
  Percentage of patients in each group requiring readmission to an acute care hospital within 30 days of discharge after an acute care hospitalization.

SECONDARY OUTCOMES:
Cause of readmissions | Up to 5 weeks
  Percentage of rehospitalizations per group for volume overload, infection or vascular access complications
Days to readmission | Up to 5 weeks
  Number of days to readmission
Average time in minutes required to perform the intervention | Up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fishbane, MD, Principal Investigator — Northshore-LIJ health system
Locations (1):
- LIJ satellite dialysis unit, Queens Village, New York, United States